CLINICAL TRIAL: NCT02711124
Title: Relationship Between Level of Glycosylated Hemoglobin and Platelet Function in Patients Undergoing Coronary Artery Bypass Grafting
Brief Title: Relationship Between Level of Hemoglobin A1c and Platelet Function in Patients Undergoing Cardiac Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Clinical Hospital Centre Zagreb (Other)
Responsible Party: Principal Investigator, Martina Zrno Mihaljević, MD, Principal Investigator, Surgeon at the Department of cardiac surgery, Clinical Hospital Centre Zagreb
Other Study IDs: KBC Zagreb
Record Dates: First submitted 2016-03-07; First posted 2016-03-17 (Estimated); Last update posted 2016-03-22 (Estimated); Status verified 2016-03

CONDITIONS: Diabetes Mellitus; Complication of Coronary Artery Bypass Graft; Blood Platelet Disorders
Keywords: hemoglobin A1c; coronary artery bypass grafting; impedance aggregometry; platelet reactivity; clinical outcomes
MeSH Terms: conditions — Diabetes Mellitus; Blood Platelet Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Group with hemoglobin A1c < 7: There will be no intervention administered to the group. The group will be observed for platelet function pre- and postoperatively.
- Group with hemoglobin A1c ≥ 7%: There will be no intervention administered to the group. The group will be observed for platelet function pre- and postoperatively.

SUMMARY:
The aim of this study is to evaluate whether increased level of hemoglobin A1c (HbA1c) correlates to higher level of platelet reactivity assessed by impedance aggregometry in patients with diabetes mellitus undergoing elective coronary artery bypass grafting (CABG).

DETAILED DESCRIPTION:
This study will be conducted at Cardiac Surgery Department, University Hospital Center Zagreb. It will be conducted in prospective observational fashion. Diabetic patients undergoing isolated, primary on-pump CABG will be consecutively recruited. Patients requiring urgent procedure will be excluded. Blood samples, both for conventional lab. findings (including HbA1c) and impedance aggregometry will be drawn prior to surgery and postoperatively on daily basis.

Cohort sample will be divided into two subgroups according to HbA1c level (Group 1 with HbA1c < 7% and Group 2 with HbA1c ≥ 7%, respectively). Respective subgroups will be compared for basic demographic data, laboratory findings including those obtained using platelet function testing, and for clinical outcomes, respectively.

Multiple-electrode aggregometry:

Whole blood aggregation will be determined using a new-generation impedance aggregometer (Multiplate analyzer; Roche Diagnostics). In brief, when platelets expose receptors on their surface they get activated and stick on the Multiplate sensor wires enhancing the electrical resistance between them. An increase in impedance is expressed in arbitrary area under the curve (AUC) units. Platelet aggregation is determined in response to stimulation with arachidonic acid (ASPI (aspirin-sensitive patients identification) test designed to evaluate the effect to acetylsalicylic acid (ASA)) and adenosine diphosphate (ADP) (ADP test designed to evaluate the effect of thienopyridines, such as clopidogrel).

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing isolated primary on-pump CABG
* Elective surgery
* Diabetic patients including insulin-dependent diabetes mellitus (IDDM) and non-insulin-dependent diabetes mellitus NIDDM
* Patients on antiplatelet therapy (aspirin and/or clopidogrel) pre- and postoperatively

Exclusion Criteria:

* Missing consent
* Patients with cardiac surgical procedures other than isolated CABG
* Patients on antiplatelet therapy other than aspirin or clopidogrel
* Urgent surgery
* Off-pump CABG
* Redo CABG

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Study population are the diabetic patients undergoing coronary artery bypass grafting at the department of cardiac surgery (The University Hospital Centre Zagreb, Croatia).
  The patients will be sampled in consecutive fashion. Cohort sample will be divided into two subgroups according to HbA1c level (Group 1 with HbA1c < 7% and Group 2 with HbA1c ≥ 7%, respectively).
Sampling Method: Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2014-02; Primary Completion 2016-08 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
The level of preoperative HbA1c that will be a predictor of the higher prevalence of platelet resistance to the aspirin | 4 days after surgery

SECONDARY OUTCOMES:
Differences in perioperative aspirin resistance (AUC, area under the curve) between patients with insulin-dependent diabetes mellitus and patients with non-insulin-dependent diabetes mellitus | 4 days after surgery
Correlation between platelet ADP receptors reactivity (AUC) and the type of diabetes | 4 days after surgery
Correlation of diabetes duration and platelet reactivity (AUC) | 4 days after surgery
The prevalence of major adverse cardiovascular events (MAACE) in patients with HbA1c ≥ 7% | 3 months after surgery
Postoperative thoracic drainage in patients with the appropriate glucose regulation (Hba1c<7%) | within the first 5 days after surgery
Mortality | 3 months after surgery
The level of HbA1c, that will represent the reliable predictor of platelet hyperreactivity and MAACE | within the 3 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Martina Zrno Mihaljević, Principal Investigator; Bojan Biočina, Study Chair; Mate Petričević, Study Director
Locations (1):
- The University Hospital Centre Zagreb, Department of cardiac surgery, Zagreb, Croatia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Thourani VH, Weintraub WS, Stein B, Gebhart SS, Craver JM, Jones EL, Guyton RA. Influence of diabetes mellitus on early and late outcome after coronary artery bypass grafting. Ann Thorac Surg. 1999 Apr;67(4):1045-52. doi: 10.1016/s0003-4975(99)00143-5. PMID 10320249
- [Background] Woods SE, Smith JM, Sohail S, Sarah A, Engle A. The influence of type 2 diabetes mellitus in patients undergoing coronary artery bypass graft surgery: an 8-year prospective cohort study. Chest. 2004 Dec;126(6):1789-95. doi: 10.1378/chest.126.6.1789. PMID 15596675
- [Background] Lazar HL, Chipkin SR, Fitzgerald CA, Bao Y, Cabral H, Apstein CS. Tight glycemic control in diabetic coronary artery bypass graft patients improves perioperative outcomes and decreases recurrent ischemic events. Circulation. 2004 Mar 30;109(12):1497-502. doi: 10.1161/01.CIR.0000121747.71054.79. Epub 2004 Mar 8. PMID 15006999
- [Background] Furnary AP, Gao G, Grunkemeier GL, Wu Y, Zerr KJ, Bookin SO, Floten HS, Starr A. Continuous insulin infusion reduces mortality in patients with diabetes undergoing coronary artery bypass grafting. J Thorac Cardiovasc Surg. 2003 May;125(5):1007-21. doi: 10.1067/mtc.2003.181. PMID 12771873
- [Background] Halkos ME, Puskas JD, Lattouf OM, Kilgo P, Kerendi F, Song HK, Guyton RA, Thourani VH. Elevated preoperative hemoglobin A1c level is predictive of adverse events after coronary artery bypass surgery. J Thorac Cardiovasc Surg. 2008 Sep;136(3):631-40. doi: 10.1016/j.jtcvs.2008.02.091. PMID 18805264
- [Background] Kempfert J, Anger K, Rastan A, Krabbes S, Lehmann S, Garbade J, Sauer M, Walther T, Dhein S, Mohr FW. Postoperative development of aspirin resistance following coronary artery bypass. Eur J Clin Invest. 2009 Sep;39(9):769-74. doi: 10.1111/j.1365-2362.2009.02175.x. PMID 19674078
- [Background] Petricevic M, Biocina B, Konosic S, Burcar I, Siric F, Mihaljevic MZ, Ivancan V, Svetina L, Gasparovic H. Definition of acetylsalicylic acid resistance using whole blood impedance aggregometry in patients undergoing coronary artery surgery. Coll Antropol. 2013 Sep;37(3):833-9. PMID 24308225
- [Background] Petricevic M, Biocina B, Konosic S, Kopjar T, Kunac N, Gasparovic H. Assessment of platelet function by whole blood impedance aggregometry in coronary artery bypass grafting patients on acetylsalicylic acid treatment may prompt a switch to dual antiplatelet therapy. Heart Vessels. 2013 Jan;28(1):57-65. doi: 10.1007/s00380-011-0216-3. Epub 2011 Dec 28. PMID 22203409